CLINICAL TRIAL: NCT00059475
Title: Randomized Comparison of Peptide Immunization in Patients at High Risk for Recurrence of Melanoma
Brief Title: Peptide Vaccination for Patients at High Risk for Recurrent Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, Dr. Steven Rosenberg, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030172; 03-C-0172; NCT00062218 (obsolete NCT alias)
Record Dates: First submitted 2003-04-26; First posted 2003-04-28 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Melanoma
Keywords: Adjuvant Therapy; MART-1 Peptides; GP100 Peptide; Immunologic Response; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Adj-2 MART-1: 27-35 (Experimental): melanoma antigen recognized by T-cells (MART)-1:27-35 peptide every three weeks for four cycles (Arm I).
  Interventions: Drug: Montanide ISA 51; Drug: Melanoma antigen recognized by T-cells (MART)-1: 27-35
- Adj-2 HD IL-2 after MART-1: 27-35 (Experimental): High-dose (HD) bolus interleukin-2 (IL-2) (720,000 IU/kg every 8 hours for up to 12 doses) after enrollment on Arm I (Arm IA)
  Interventions: Drug: Interleukin-2 (IL-2); Drug: Montanide ISA 51; Drug: Melanoma antigen recognized by T-cells (MART)-1: 27-35
- Adj-2 27-35 (27L) MART-1 (Mod9mer) peptide Q3wks x 4 (Experimental): 27-35(27L):melanoma antigen recognized by T-cells (MART)-1 peptide every three weeks for four cycles (Arm II).
  Interventions: Drug: Montanide ISA 51; Drug: 27-35 (27L): melanoma antigen recognized by T-cells (MART)-1
- Adj-2 HD IL-2 after 27-35 (27L): MART-1 (Mod9mer) (Experimental): High-dose (HD) bolus interleukin-2 (IL-2) (720,000 IU/kg every 8 hours for up to 12 doses) after enrollment on Arm II (Arm IIA)
  Interventions: Drug: Interleukin-2 (IL-2); Drug: Montanide ISA 51; Drug: 27-35 (27L): melanoma antigen recognized by T-cells (MART)-1
- Adj-2 MART-1: 26-35 (27L) (Mod10mer) peptide Q3wks x 4 (Experimental): melanoma antigen recognized by T-cells (MART)-1:26-35(27L) peptide every three weeks for four cycles (Arm III).
  Interventions: Drug: Montanide ISA 51; Drug: melanoma antigen recognized by T-cells (MART)-1: 26-35(27L)
- Adj-2 HD IL-2 after MART-1: 26-35 (27L) (Mod10mer) (Experimental): High-dose (HD) bolus interleukin-2 (IL-2) (720,000 IU/kg every 8 hours for up to 12 doses) after enrollment on Arm III (Arm IIIA)
  Interventions: Drug: Interleukin-2 (IL-2); Drug: Montanide ISA 51; Drug: melanoma antigen recognized by T-cells (MART)-1: 26-35(27L)
- Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 (Experimental): 27-35(27L):melanoma antigen recognized by T-cells (MART)-1 peptide plus the gp100:209-217(210M) peptide emulsified together every three weeks for four cycles (Arm IV).
  Interventions: Drug: Glycoprotein 100 (GP100): 209-217 (210M); Drug: Montanide ISA 51; Drug: 27-35 (27L): melanoma antigen recognized by T-cells (MART)-1
- Adj-2 HD IL-2 after 27-35 (27L): MART-1 + gp209-2M (Experimental): High-dose (HD) bolus interleukin-2 (IL-2) (720,000 IU/kg every 8 hours for up to 12 doses) after enrollment on Arm IV (Arm IVA)
  Interventions: Drug: Interleukin-2 (IL-2); Drug: Montanide ISA 51; Drug: 27-35 (27L): melanoma antigen recognized by T-cells (MART)-1

INTERVENTIONS:
Drug: Glycoprotein 100 (GP100): 209-217 (210M)
  Arms: Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4
Drug: Interleukin-2 (IL-2) — 720,000 IU/kg as an intravenous bolus over a 15 minute period every 8 hours and continuing for up to 4 days (a maximum of 12 doses).
  Other Names: Interleukin-2
  Arms: Adj-2 HD IL-2 after 27-35 (27L): MART-1 (Mod9mer); Adj-2 HD IL-2 after 27-35 (27L): MART-1 + gp209-2M; Adj-2 HD IL-2 after MART-1: 26-35 (27L) (Mod10mer); Adj-2 HD IL-2 after MART-1: 27-35
Drug: Montanide ISA 51
Drug: Melanoma antigen recognized by T-cells (MART)-1: 27-35
  Arms: Adj-2 HD IL-2 after MART-1: 27-35; Adj-2 MART-1: 27-35
Drug: 27-35 (27L): melanoma antigen recognized by T-cells (MART)-1
  Arms: Adj-2 27-35 (27L) MART-1 (Mod9mer) peptide Q3wks x 4; Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4; Adj-2 HD IL-2 after 27-35 (27L): MART-1 (Mod9mer); Adj-2 HD IL-2 after 27-35 (27L): MART-1 + gp209-2M
Drug: melanoma antigen recognized by T-cells (MART)-1: 26-35(27L)
  Arms: Adj-2 HD IL-2 after MART-1: 26-35 (27L) (Mod10mer); Adj-2 MART-1: 26-35 (27L) (Mod10mer) peptide Q3wks x 4

SUMMARY:
This study will examine the effectiveness and side effects of an experimental vaccine to prevent recurrence of melanoma. The likelihood of melanoma returning is higher in patients who have melanoma lesions deep in the skin, in patients who have had positive lymph nodes, and in patients who have had surgery for metastatic disease (cancer that has spread beyond the primary site). Melanoma tumors produce proteins called glycoprotein 100 (gp100) and melanoma-associated antigen recognized by T cells 1 (MART-1). Vaccination with specific pieces of these proteins (peptides) may boost the immune system's fight against the cancer. The vaccine injections are mixed with an oil-based substance called Montanide ISA-51, which is intended to increase the immune response to the peptide.

Patients 16 years of age and older whose melanoma has been surgically removed and who are currently free of disease may be eligible for this study. Candidates will be screened with a physical examination and blood and urine tests. An electrocardiogram (EKG), x-rays and other imaging studies will be done if recent results are not available. Some candidates may require heart tests, such as a cardiac stress test or echocardiogram, or lung function tests. In addition, all candidates will be tested for human leukocyte antigen (HLA) tissue type; patients must be type human leukocyte antigens (HLA-A)*0201, the type on which this vaccine is based.

Participants will be randomly assigned to receive one of four different vaccines to determine which peptides offer the best immunity. Each treatment course consists of two injections of the vaccines every 3 weeks for four times. The injections are given under the skin of the thigh. After every other treatment course (every 6 months), patients will undergo a series of x-rays and scans to look for tumor. The immunizations may continue for up to 12 months as long as the melanoma does not return. The injections are given at the National Institutes of Health (NIH) Clinical Center. Patients are monitored for 1 hour after each injection and have blood tests and a physical examination to look for treatment side effects.

Patients will be followed with blood tests every 12 weeks to monitor body functions. They will also undergo leukapheresis-a procedure to collect white blood cells-before starting treatment and about 3 to 4 weeks after the fourth vaccine to evaluate how the vaccines affect the action of the immune system cells. For this procedure, blood is drawn through a needle in the arm, similar to donating blood. The blood goes through a machine that separates out the lymphocytes (white blood cells), and the rest of the blood is returned through a needle in the other arm. Some patients may undergo a biopsy-surgical removal of a small piece of tissue under local anesthetic-of normal skin and tumor or lymph node tissue to examine the effects of the vaccines on the tumor immune cells.

Patients whose disease returns during the first course of vaccine therapy will have surgery to remove the tumor and will continue to receive the vaccine treatment. Patients whose tumor returns after completing one course of therapy may receive a substance called interleukin-2 (IL-2), which can boost immune function against the tumor. interleukin-2 (IL-2) is given intravenously (through a small tube placed in a vein) every 8 hours for 4 days. This regimen is repeated after 10 to 14 days. Those who respond to interleukin-2 (IL-2) will have a third course of treatment after 2 months. Patients whose disease recurs after treatment will be taken off the study and will be referred back to their referring physician or to another study, if an appropriate one is available.

DETAILED DESCRIPTION:
Human leukocyte antigens (HLA-A)*0201 positive patients at high risk for recurrence of melanoma, or completely resected metastatic melanoma will receive immunization with peptides representing human leukocyte antigen (HLA)-restricted T cell epitopes of the melanoma antigen recognized by T-cells (MART-1) or glycoprotein 100 (gp100) melanoma antigens emulsified in Montanide ISA-51 or Montanide trademark(TM) ISA 51 vegetable grade (VG). Patients will be randomized to receive one of three different melanoma antigen recognized by T-cells (MART-1) peptides or to receive a combination of a melanoma antigen recognized by T-cells (MART-1) peptide plus a glycoprotein 100 (gp100) peptide. This study is designed to evaluate the immunologic effects of the different peptide immunizations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Human leukocyte antigens (HLA-A)*0201 patients, age greater than or equal to 16 years, with lesions greater than or equal to 1.5 mm in thickness, or greater than or equal to 1 positive lymph node, or ulcerated lesions, or local recurrence, or completely resected metastatic melanoma, within 6 months of surgical resection will be considered. Patients must be clinically disease free at the time of protocol entry as documented by radiologic studies within 6 weeks of patient entry.

Serum creatinine of 2.0 mg/dl or less.

Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

White blood cell (WBC) 3000/mm^3 or greater.

Platelet count 90,000 mm^3 or greater.

Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than three times normal.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Patients of both genders must be willing to practice effective birth control during this trial because the potential for teratogenic effects are unknown.

Patients may have had prior adjuvant treatment with immunotherapy, including interferon, or may have had treatment for metastatic disease and are now no evidence of disease (NED), including chemotherapy or biotherapy, as long as 3 weeks have elapsed since prior systemic therapy.

EXCLUSION CRITERIA:

Patients will be excluded:

1. who have ocular or mucosal melanoma.
2. who are undergoing or have undergone in the past 3 weeks any systemic therapy except surgery for their cancer, and must have recovered from any adverse effects of treatment prior to entry, other than those that do not have clinical implications, e.g. vitiligo, alopecia.
3. have active systemic infections, autoimmune disease or any known immunodeficiency disease.
4. who require systemic steroid therapy.
5. who are pregnant or breastfeeding.
6. who are known to be positive for hepatitis B surface antigen (B(s)AG) or human immunodeficiency virus (HIV) antibody.
7. who have any form of active primary or secondary immunodeficiency or who have not recovered immune competence after chemotherapy or radiation therapy.
8. who have previously been immunized with melanoma antigen recognized by T-cells (MART)-1.
9. who have known hypersensitivity to any of the agents used in this study.

ELIGIBILITY FOR ADMINISTRATION OF Interleukin-2 (IL-2):

Patients who develop progressive disease while receiving peptide alone must meet the following criteria to be eligible to receive Interleukin-2 (IL-2):

1. Patients must have measurable metastatic melanoma.
2. Patients may not have active major medical illnesses such as cardiac ischemia, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Patients with recent prolonged history of cigarette smoking or symptoms of respiratory dysfunction must have a normal pulmonary function test as evidenced by a forced expiratory volume 1 (FEV 1) greater than 60% predicted.
4. Patients with electrocardiogam (EKG) abnormalities, symptoms of cardiac ischemia or arrhythmias or age greater than 50 years will have a normal stress cardiac test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine echocardiogram or other stress test).
5. Patients must be willing to sign a durable power of attorney (DPA).
6. Serum creatinine of 2.0 mg/dl or less.
7. Total bilirubin 2.0 mg/dl or less, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
8. White blood cell (WBC) 3000/mm^3 or greater.
9. Platelet count 90,000 mm^3 or greater.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2003-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2003-C-0172.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were accrued to this trial.
Period: Overall Study
Arm/Group | Adj-2 MART-1: 27-35 | Adj-2 HD IL-2 After MART-1: 27-35 | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M
Started | 33 | 2 | 24 | 3 | 33 | 2 | 34 | 7
Completed | 33 | 2 | 24 | 3 | 33 | 2 | 34 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adj-2 MART-1: 27-35 | Adj-2 HD IL-2 After MART-1: 27-35 | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M | Total
Number analyzed (Participants) | 33 | 2 | 24 | 3 | 33 | 2 | 34 | 7 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 30 | 2 | 20 | 3 | 29 | 2 | 33 | 7 | 126
  >=65 years | 3 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (14.9) | 42.0 (8.5) | 48.5 (12.9) | 52.7 (3.8) | 47.5 (13.0) | 52.0 (8.5) | 44.9 (11.4) | 48.0 (8.5) | 47.55 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 6 | 0 | 14 | 0 | 15 | 4 | 54
  Male | 20 | 0 | 18 | 3 | 19 | 2 | 19 | 3 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 33 | 2 | 24 | 3 | 32 | 2 | 34 | 7 | 137
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 33 | 2 | 23 | 3 | 33 | 2 | 34 | 7 | 137
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 2 | 24 | 3 | 33 | 2 | 34 | 7 | 138

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Response Rate
Description: Immunologic monitoring will be conducted using in vitro sensitization assays. The immunologic response in these assays will be considered positive if at least a two-fold increase in vaccine specific interferon gamma (y-IFN) secretion is seen between post vaccination specimens compared to the pre vaccination specimens.
Time Frame: 11 months
Population: The number of participants analyzed and results are correct. We do not have the immunologic response rate data for all patients.
Measure: Number; unit: Participants
Arm/Group | Adj-2 MART-1: 27-35 | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4
Number analyzed (Participants) | 13 | 13 | 13 | 8
Participants | 7 | 1 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For details about the adverse events see the adverse event module.
Time Frame: 11 months
Measure: Number; unit: Participants
Arm/Group | Adj-2 MART-1: 27-35 | Adj-2 HD IL-2 After MART-1: 27-35 | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M
Number analyzed (Participants) | 33 | 2 | 24 | 3 | 33 | 2 | 34 | 7
Participants | 31 | 2 | 20 | 3 | 32 | 2 | 30 | 7

3. Primary Outcome: Response Rate
Description: Response is measured from the time measurement criteria are first met for complete response (CR) or partial response (PR) (whichever is first) until the first date that recurrent disease is objectively documented. Complete response is the disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: 6 years
Population: The number of participants analyzed and results are correct. We do not have the response rate data for all patients.
Measure: Number; unit: participants
Arm/Group | Adj-2 HD IL-2 After MART-1: 27-35 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M
Number analyzed (Participants) | 2 | 3 | 2 | 7
participants | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Adj-2 MART-1: 27-35 | Adj-2 HD IL-2 After MART-1: 27-35 | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/2 | 0/24 | 0/3 | 0/33 | 1/2 | 0/34 | 0/7
Other Adverse Events (participants affected / at risk) | 31/33 | 2/2 | 20/24 | 3/3 | 32/33 | 2/2 | 30/34 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adj-2 MART-1: 27-35 (N=33) | Adj-2 HD IL-2 After MART-1: 27-35 (N=2) | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 (N=24) | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) (N=3) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 (N=33) | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) (N=2) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 (N=34) | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M (N=7)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adj-2 MART-1: 27-35 (N=33) | Adj-2 HD IL-2 After MART-1: 27-35 (N=2) | Adj-2 27-35 (27L) MART-1 (Mod9mer) Peptide Q3wks x 4 (N=24) | Adj-2 HD IL-2 After 27-35 (27L): MART-1 (Mod9mer) (N=3) | Adj-2 MART-1: 26-35 (27L) (Mod10mer) Peptide Q3wks x 4 (N=33) | Adj-2 HD IL-2 After MART-1: 26-35 (27L) (Mod10mer) (N=2) | Adj-2 27-35 (27L): MART-1 + gp100: 209-217 (210M) Q3wks x 4 (N=34) | Adj-2 HD IL-2 After 27-35 (27L): MART-1 + gp209-2M (N=7)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 4 (5) | 4 (5)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 31 (90) | 0 (0) | 20 (66) | 0 (0) | 32 (94) | 0 (0) | 29 (89) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 5 (6) | 0 (0) | 7 (8) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anticipated Dose Limiting Toxicity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low urine output (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No